CLINICAL TRIAL: NCT01466634
Title: Bioabsorbable Versus Permanent Polymer Bare Metal Stents in Saphenous Vein Graft Disease: Insights From a Meta-analysis of 6221 Patients
Brief Title: Bioabsorbable Versus Durable Polymer Drug Eluting Stent (DES): a Meta-analysis
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Lupi Alessandro, Dr, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: 010101
Record Dates: First submitted 2011-10-24; First posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Restenosis; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Percutaneous Coronary Intervention; Stents

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- permanent polymer DES
  Interventions: Procedure: percutaneous coronary intervention with stent
- bioabsorbable polymer DES
  Interventions: Procedure: percutaneous coronary intervention with stent

INTERVENTIONS:
Procedure: percutaneous coronary intervention with stent — patients with coronary artery disease treated by percutaneous coronary intervention with BP-DES are compared with patients with coronary artery disease treated by percutaneous coronary intervention with PP-DES

SUMMARY:
Evidence supporting use of bioabsorbable polymer drug eluting stents (BP-DES) is uncertain. Thus the investigators planned a meta-analysis to compare outcomes of BP-DES versus PP-DES in obstructive coronary artery disease.

DETAILED DESCRIPTION:
Evidence supporting use of bioabsorbable polymer drug eluting stents (BP-DES) is uncertain. Previous studies suggested that BP-DES are at least as effective as durable polymer drug eluting stents (PP-DES). Thus the investigators planned a meta-analysis to compare outcomes of BP-DES versus PP-DES in obstructive coronary artery disease. Medline and Web databases were searched for studies comparing BP-DES and PP-DES for obstructive coronary disease, reporting rates of overall mortality, target lesion revascularization (TLR), myocardial infarction (MI), binary restenosis and late lumen loss (LLL) with a follow-up ≥ 6 months. Odds ratios (ORs) will be computed from individual studies and pooled according to a fixed effect (e.g. inverse variance weighting) or random effect model in case of statistical heterogeneity. Given the a priori heterogeneous nature of the observational analyses, separate subgroup analysis of studies with PLA bioabsorbable polymer loaded with biolimus A19 (BP-BES) is prespecified.

ELIGIBILITY:
Inclusion Criteria:

* randomized studies
* studies reporting clinical outcomes as overall death and/or acute myocardial infarction and/or late stent thrombosis (ARC definition)[**] and/or target lesion revascularization and/or late lumen loss
* follow up period longer than 6 months.

Exclusion Criteria:

* duplicate reporting (in which case the manuscript reporting the largest sample or the longest follow-up was selected)
* inability to compute risk estimates due to absence of clinical event in one of the groups
* studies presenting composite major adverse cardiac event (MACE) and not individual end points.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease with indication to percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 6221 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
late coronary lumen loss | 9 month
target lesion revascularization | 9 month
overall mortality | 1 year
Late stent thrombosis | 1 year
Myocardial Infarction | 1 year

SECONDARY OUTCOMES:
Binary restenosis | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Lupi, MD, Principal Investigator — AOU Maggiore della Carita
Locations (1):
- Ospedale Maggiore della Carità, Novara, Italy

REFERENCES:
- [Derived] Lupi A, Rognoni A, Secco GG, Lazzero M, Nardi F, Fattori R, Bongo AS, Agostoni P, Sheiban I. Biodegradable versus durable polymer drug eluting stents in coronary artery disease: insights from a meta-analysis of 5,834 patients. Eur J Prev Cardiol. 2014 Apr;21(4):411-24. doi: 10.1177/2047487312467745. Epub 2012 Nov 14. PMID 23152364